CLINICAL TRIAL: NCT02082457
Title: Multi-center, Randomized, Double Blinded, Placebo-controlled, Phase II Trial to Assess the Efficacy and Safety of YKP10811 in Subjects With Irritable Bowel Syndrome With Constipation
Brief Title: Efficacy and Safety of YKP10811 in Subjects With Irritable Bowel Syndrome With Constipation
Acronym: YKP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YKP10811_IBS_II_2013
Record Dates: First submitted 2014-02-10; First posted 2014-03-10 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Irritable Bowel Syndrome; Constipation
Keywords: Irritable Bowel Syndrome; Constipation; C-IBS
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation | interventions — carbamic acid 3-(4-((4-amino-5-chloro-2-methoxybenzoylamino)methyl)piperidin-1-yl)-1-(4-fluorophenyl)propyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Two tablets of YKP10811 placebo are administered orally once a day for 12 weeks.
  Interventions: Drug: YKP10811 placebo
- YKP10811 10mg (Experimental): Two tablets of YKP10811 5mg are administered orally once a day for 12 weeks.
  Interventions: Drug: YKP10811 5mg
- YKP10811 20mg (Experimental): One tablet of YKP10811 20mg and one tablet of placebo are administered orally once a day for 12 weeks.
  Interventions: Drug: YKP10811 20mg; Drug: YKP10811 placebo
- YKP10811 40mg (Experimental): Two tablets of YKP10811 20mg are administered orally once a day for 12 weeks.
  Interventions: Drug: YKP10811 20mg

INTERVENTIONS:
Drug: YKP10811 5mg
  Arms: YKP10811 10mg
Drug: YKP10811 20mg
  Arms: YKP10811 20mg; YKP10811 40mg
Drug: YKP10811 placebo
  Arms: Placebo; YKP10811 20mg

SUMMARY:
This trial is to investigate efficacy and safety of YKP10811 in Subjects With Irritable Bowel Syndrome With Constipation. The difference of responder rate between test group (10, 20 and 40mg) and placebo will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. more than 18 years old
2. patients met with ROME III criteria for C-type IBS

Exclusion Criteria:

* pregnancy or lactation
* a history of surgery for gastrointestinal tract
* a history of gastrointestinal bleeding, diverticulitis and ileus within 1 year of screening visit
* inflammatory bowel disease or malignant tumor within 5 years of screening visit
* taking drugs that could have impact on efficacy assessment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Abdominal pain intensity & stool frequency responder | 12weeks
  an improvement of equl and more than 30% from baseline in the average of the daily worst abdominal pain score and an increase of equal and more than 1 CSBM from baseline

SECONDARY OUTCOMES:
subject global assessment | 12 weeks
  the degree of symptom relief on abdominal pain, bloating, stool frequency, stool consistency, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Hyo jin Park, MD.PhD., Principal Investigator — Gang Nam Severance Hospital
Locations (1):
- Gang Nam Severance Hospital, Gang Nam Gu, Seoul, South Korea